CLINICAL TRIAL: NCT03609541
Title: Evaluation of Biomarkers of COPD Exacerbation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Daniela Gompelmann, PD Dr. med. Daniela Gompelmann, Heidelberg University
Other Study IDs: Protocol DG2.0-08.05.2018
Record Dates: First submitted 2018-07-16; First posted 2018-08-01 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: SAA Level and SAA/Lipoxin A4 Ratio

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with stable COPD: Evaluation of serum amlyoid A, lipoxin A4, CRP and fibrinogen
- Patient with COPD exacerbation: Evaluation of serum amlyoid A, lipoxin A4, CRP and Fibrinogen at beginning and at the end of COPD exacerbation

SUMMARY:
Serum amlyoid A (SAA) was shown to act as biomarker for exacerbation of chronic obstructive pulmonary disease (AE-COPD). It seems that SAA triggers chronic inflammation by binding to ALX/PFR2 receptor. In contrast, lipoxin A4 seems to inhibit the inflammatory processes by binding to ALX/PFR2 receptor. A small trial has already demonstrated an imbalance between SAA and lipoxin A4 during AE-COPD. This study evaluates SAA level and SAA/lipoxin A4 ratio in patients with stable COPD and AE-COPD.

DETAILED DESCRIPTION:
Patient enrolment and data aquisition is to be carried out on a prospective basis. It is planned to enrol 40 patients with stable COPD and 40 patients with AE-COPD. All patients will undergo blood sampling inlcuding SAA and Lipoxin A4.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD GOLD 3-4 confirmed by anamnesis and pulmonary function test
* Patient has provided written informed consent

Exclusion Criteria:

* other reasons for worsening of symptoms (cough, dyspnea): e.g. pneumothorax, pneumonia, pulmonary embolism, myocardial infarction.
* malignant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD GOLD 3-4 confirmed by anamnesis and pulmonary function test (stable COPD and COPD exacerbation)
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
SAA | time of exacerbation/hospitalisation, an average of 3 days
  SAA level in stable COPD and COPD exacerbation
SAA/lipoxin A4 ratio | time of exacerbation/hospitalisation, an average of 3 days
  SAA/lipoxin A4 ratio in stable COPD and COPD exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Gompelmann, MD, Principal Investigator — Thoraxklinik University of Heidelberg
Locations (1):
- Thoraxklinik Heidelberg, Heidelberg, Germany